CLINICAL TRIAL: NCT02864134
Title: Predictive Effect of Ganglion Cell Layer on Visual Acuity at 6 Months and on Visual Function at 1 Year After an Episode of Optic Neuritis
Brief Title: Optic Neuritis and Ganglion Cell Layer
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Andréane Lavallée, Ophthalmologist, CHU de Quebec-Universite Laval
Other Study IDs: 2017-2916
Record Dates: First submitted 2016-08-05; First posted 2016-08-11 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Optic Neuritis
Keywords: Optic neuritis; ganglion cell layer
MeSH Terms: conditions — Optic Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
BACKGROUND AND OBJECTIVES: The recent expansion of the applications of optical coherence tomography (OCT) demonstrated a higher correlation between the analysis of ganglion cells and visual function, in comparison with the analysis of the nerve fiber layer for several diseases of the optic nerve. Atrophy of the ganglion cells tends to induce the visual function deficits. In the case of optic neuritis, inflammation of the optic nerve causes a deficit of visual function initially with low vision, color blindness and visual field. Secondary atrophy of ganglion cell can result. The purpose of the study is to evaluate the correlation between the analysis of ganglion cells at the time of diagnosis of optic neuritis and the resulting visual acuity at 6 months and visual function (visual acuity, color vision and perimetry) 1 year regardless of treatment. A predictive effect could help predict the patient's clinical course and management of uncertainty and anxiety. MATERIALS AND METHODS: An assessment at diagnosis and follow-ups at 6 months and 1 year with a measurement of best corrected visual acuity, a test color vision HRR (Hardy-Rand-Rittler), an OCT with analysis of ganglion cells and perimetry Humphrey 30 -2 fast will be done. Simple linear and logistic regressions will be used. RESULTS: We expect that there will be a significant association between atrophy of ganglion cells in the diagnosis and residual visual function after an episode of optic neuritis. We believe that the initial atrophy is associated with poorer visual prognosis. CONCLUSION: A predictive effect could help to inform the patient about the evolution of the disease and provide early visual rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Major and apt patients seen in consultation with diagnosis of optic neuritis

Exclusion Criteria:

* Concomitant ophthalmic diseases

  * known macular pathology
  * Amblyopia
  * Glaucoma
  * History of an ophthalmic surgery
  * Family history of hereditary optic neuropathy
  * Pathological myopia (refractive error of 8 diopters or more).
* Known neurological disease other than multiple sclerosis.
* Habit

  * Nutritional deficiency anorexia, restrictive gastrointestinal surgery.
* Active or former professional or recreational exposure

  * Exposure to metals: lead, mercury, thallium
  * Exposure to solvents: ethylene glycol, toluene, styrene, perchlorethylene;
  * Prior poisoning: methanol, carbon dioxide.
* Usual or earlier Medication

  * Taking one or more drugs known to cause toxic optic neuropathy*

    * listed available on demand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major and apt patients seen in consultation with diagnosis of optic neuritis in emergency context
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-08; Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Association between the analysis of ganglion cells at diagnosis and the resulting visual acuity at 6 months after optic neuritis | 6 months post optic neuritis
  Evaluation of best corrected visual acuity at 6 months post optic neuritis episode in correlation with initial ganglion cell layer analysis measures in order to predict the visual acuity in the future.
Association between the analysis of ganglion cells at diagnosis and the visual function at 12 months after optic neuritis | 12 months post optic neuritis
  Evaluation of the visual function (best corrected visual acuity, perimetry, color vision) at 12 months post optic neuritis episode in correlation with initial ganglion cell layer analysis measures in order to predict the visual acuity in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Andréane Lavallée, MD, FRCSC, Principal Investigator — CHU de Québec-Laval University
Locations (1):
- Hopital Saint-Sacrement, Québec, Canada

IPD SHARING:
Plan to Share IPD: No